CLINICAL TRIAL: NCT05045950
Title: Optimizing Neurocognition With Whole Brain Radiation Therapy (WBRT) Using Upfront Pulsed Reduced Dose-Rate (PRDR) Technique (ONCO-RT) - A Phase II Trial of Upfront Pulsed Reduced Dose Rate Whole-Brain Radiation Therapy for Brain Metastases
Brief Title: Optimizing Neurocognition With Whole Brain Radiation Therapy (WBRT) Using Upfront Pulsed Reduced Dose-Rate (PRDR) Technique
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Lindsay Puckett, MD, Assistant Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00041354
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Brain Metastases
Keywords: whole-brain radiation therapy; upfront pulsed reduced dose-rate
MeSH Terms: conditions — Brain Neoplasms | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- WBRT-PRDR plus memantine. (Experimental): Study patients will receive WBRT-PRDR within 14 days of registration. All patients will receive single daily fractions using 3D conformal radiotherapy. A dose of 30 Gy in 10 fractions will be delivered using the PRDR technique. Memantine should ideally start two days (or one day) prior to WBRT PRDR and must start no later than the fourth WBRT PRDR treatment and will continue for a maximum of 24 weeks (≈six months). Memantine will be administered as per standard institutional guidelines.
  Interventions: Drug: Memantine -Twice Daily or Extended Release; Radiation: WBRT utilizing the PRDR technique

INTERVENTIONS:
Drug: Memantine -Twice Daily or Extended Release — Both extended release memantine and twice daily memantine dosing will be allowed.
  Twice daily dosing:
  The target dose for memantine is 20 mg (10 mg divided twice daily). Dose will be escalated by 5 mg each week to a target of 10 mg twice daily (i.e., 5 mg a day on week 1, then 5 mg twice daily (BID) on week 2, then 10 mg in AM plus 5 mg in PM on week 3, followed by 10 mg in AM plus 10 mg in PM by week 4).
  Extended Release Memantine:
  The target dose for extended release memantine is 28 mg. Dose will be escalated by 7 mg per week to a target of 28 mg daily (i.e., 7 mg a day on week 1, then 14 mg a day on week 2, then 21 mg a day on week 3, followed by 28 mg a day by week 4).
  Other Names: Namenda
Radiation: WBRT utilizing the PRDR technique — The total dose of 3000 cGy (30 Gy) will be divided 10 fractions of 300 cGy (3 Gy); each fraction will be delivered as a series of 20 cGy (0.2Gy) pulses separated by 3 min time intervals. 20 cGy / 3 min = 6.67 cGy/min (or 0.0667 Gy/min). Total time is determined by the fractionated series and time intervals, meaning 300cGy/20cGy = 15 division x 3 minutes = 45 minutes. Including time to set up, approximate total time per treatment session will be 60 minutes.

SUMMARY:
Study patients will receive Whole-brain radiation therapy (WBRT) - pulsed reduced dose rate (PRDR) within 14 days of registration. All patients will receive single daily fractions using 3D conformal radiotherapy. A dose of 30 Gy in 10 fractions will be delivered using the PRDR technique.

DETAILED DESCRIPTION:
This is a phase II, single-arm, multi-center study assessing the feasibility and tolerance of WBRT using upfront PRDR in the treatment of solid tumor brain metastases. This study will also examine the impact of substituting PRDR for standard whole-brain radiation therapy in the upfront treatment of brain metastases on neurocognitive decline as compared to historical controls. Additionally, clinical patient outcomes associated with radiation treatment of brain metastases will be collected. Using a group sequential design with one interim analysis to stop for futility, the investigators will recruit and enroll 53 adult patients (≥18 years) undergoing upfront treatment of brain metastases to determine feasibility and a preliminary analysis after the first 27 enrolled patients.

In order to be eligible for this study, patients must have a biopsy-proven solid malignancy with intracranial lesions radiographically consistent with or pathologically proven to be brain metastases. Patient who are confirmed to meet all eligibility criteria will be registered to the study and start PRDR WBRT within two weeks postregistration. Patients will receive PRDR WBRT as a dose of 30Gy in 10 fractions and start memantine orally two days prior to (or one day prior to) but no later than the fourth PRDR WBRT treatment session.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at diagnosis of brain metastases.
2. Eastern Cooperative Oncology Group (ECOG) Performance Score of <2.
3. Participants must have a biopsy-proven solid malignancy (histologic proof or unequivocal cytologic proof solid tumor malignancy from either the primary or any metastatic site) with intracranial lesions radiographically consistent with or pathologically proven to be brain metastases.
4. Patients who have undergone prior systemic therapy are eligible.
5. Life expectancy from extracranial disease greater than six months.
6. Patients with measurable brain metastasis.
7. Patients may have had prior therapy for brain metastasis, including stereotactic radiosurgery (SRS)and surgical resection. Patients must have completed prior therapy by at least 7 days prior to study enrollment for SRS and at least 14 days for surgical resection
8. If an open biopsy is performed, the patient must be at least one-week post-biopsy. This requirement is not necessary for stereotactic biopsies.
9. Creatinine clearance is ≥ 30 mL/min.
10. Start of PRDR WBRT within two weeks following registration.
11. Ability to complete the Neurocognitive Function (NCF) test battery (including people whose primary language is English).
12. Patients with previous or other malignancies whose disease is controlled and not impacting ECOG performance or life expectancy.
13. Willing and able to give consent and to comply with treatment and follow-up schedule.

Exclusion Criteria:

1. Metastases from hematological malignancy, or central nervous system malignancy.
2. Patients whose malignancy is being treated with curative intent.
3. Leptomeningeal metastases.
4. Contraindication to MRI imaging with contrast.
5. Contraindication to memantine including concurrent use of N-methyl-D-aspartate (NMDA) antagonists.
6. Stage IV-V chronic kidney disease or end-stage renal disease.
7. Participants with a maximum tumor diameter exceeding 5 cm (if not resected).
8. Prior cranial whole brain radiation therapy.
9. Past medical history of dementia which is thought to be unrelated to the brain metastases.
10. Women of childbearing potential who are known to be pregnant or are unwilling to use an acceptable method of contraception from the time of informed consent until completion of the course of radiotherapy.
11. Patients must not have a serious medical or psychiatric illness that would, in the opinion of the treating physician, prevent informed consent or completion of protocol treatment, and/or follow-up visits.
12. Non-native English speakers will be excluded since patients often lose their faculty with the language they acquired second before their native language is affected in the context of cognitive decline. This could adversely affect performance on verbal cognitive tasks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Successful completion of PRDR WBRT treatment | 5 days
  The number of subjects successfully completing PRDR WBRT treatment within five days of intended treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Puckett, MD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Clement J. Zablocki Veterans Affairs Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No